CLINICAL TRIAL: NCT05000853
Title: New Pathophysiological Pathways Involved in Iron Metabolism Disorder in Heart Failure: The IRON-PATH II Investigator Initiated Study
Brief Title: New Pathophysiological Pathways Involved in Iron Metabolism Disorder in Heart Failure
Acronym: IRON-PATH II
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Josep Comín, Prof. Josep Comín-Colet, MD, PhD, Hospital Universitari de Bellvitge
Other Study IDs: IDIBELL - EOM019/21
Record Dates: First submitted 2021-07-15; First posted 2021-08-11 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Heart Failure
Keywords: Iron Deficiency; Machine Learning; Multi-Omics Approaches; Outcomes Research
MeSH Terms: conditions — Heart Failure; Iron Deficiencies | interventions — ferric carboxymaltose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with iron deficiency
  Interventions: Drug: Iron Carboxymaltose
- Patients without iron deficiency

INTERVENTIONS:
Drug: Iron Carboxymaltose — Iron supplementation when is needed according to usual care
  Groups: Patients with iron deficiency

SUMMARY:
The aim of our study is to understand the biological pathways involved in the occurrence of IDy in patients with HF since ID is very common and supposes a negative impact in terms of clinical outcomes in these patients. In this context, a deeper understanding of the mechanisms involved in the development of ID in these patients and the impact on the altered biological pathways after iron replenishment will pave the way for an improvement and simplification of the preventive strategies in patients with HF.

DETAILED DESCRIPTION:
The IRON-PATH II Project is a pre-clinical and clinical study designed as a multicenter, prospective, observational (non-interventional), investigator initiated study. The total number of patients to be recruited will be 210 (80 patients without ID and 130 patients with ID). Patients will be recruited during 12 months in 7 centers across Spain and Portugal and followed for a fixed period of 12 months. The primary objective of the clinical study is to define pathways associated with systemic and tissue ID in HF patients compared with non-ID HF patients and explore the change in the patterns of pathway activation/suppression after irons status normalization in ID patients with intravenous iron treatment using an integrative omics and systems biology approach including whole-genome analysis of gene expression (transcriptome), protein synthesis (proteomics) and metabolic characterization (metabolomics) from blood samples. Key secondary objectives will include changes in patient-reported outcomes (PROMs) such as QoL, patient-reported experience measures (PREMs), the occurrence of events, among others between those with and without ID. The aims of the pre-clinical study is to confirm previous findings of the IRONPATH I study and to explore in vitro interventions in cardiac cells models with iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* HF diagnosis according to European Society of Cardiology
* LVEF≤50% (systolic HF).
* Patients receiving oral standard medication for chronic HF.
* Iron status evaluated in the last 3 months.
* Written informed consent.

Exclusion Criteria:

* Age<18 years old.
* Intravenous or oral iron administration or under treatment with ESA (erythropoiesis-stimulating agents) in the previous 3 months.
* Planned cardiac resynchronization therapy (CRT), revascularization and other major interventions including heart transplant or left ventricular assist device (LVAD) implantation in the next 3 months in patients with ID.
* Planned uptitration of guideline-mandatory HF-modifying drugs in the next 3 months (except iron repletion) in patients with ID.
* Moderate or severe anaemia (Hb<11 g/dL).
* The patient is unable or unwilling to give the informed consent to participate.
* Unstable patients with signs of fluid overload or low cardiac output at the moment of enrollment.
* Life expectancy less than 1 year (excluding HF).
* The patient is considered not to be an adequate candidate for this study according to the decision of the local investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort will be a multicenter, observational, prospective, cross-sectional and longitudinal nested case-control sample of 210 patients with (130 cases) and without (80 controls) ID according to the FAIR-HF (27) (serum ferritin <100 mg/L or transferrin saturation [%TSAT]<20% if ferritin is between 100-300mg/L), recruited for the specific purpose of the IRON-PATH II study.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
To define pathways associated with iron deficiency (ID) in heart failure (HF) patients compared with non-ID HF patients | Twelve months after inclusion the patient
  Using an integrative omics and systems biology approach including whole-genome analysis of gene expression (transcriptome), protein synthesis (proteomics) and metabolic characterization (metabolomics) from blood samples.

SECONDARY OUTCOMES:
Functional Biomarkers (New York Heart Association [NYHA) | Twelve months after inclusion the patient
  Comparison between ID and non ID patients
Improvement of self-care using a validated scale (European Heart Failure Self-Care Behavior Scale). | Twelve months after inclusion the patient
  Comparison between ID and non ID patients
Patient-reported experience measures (PREMs) (IEXPAC) | Twelve months after inclusion the patient
  Comparison between ID and non ID patients
Prognostic biomarkers (NT-proBNP) | Twelve months after inclusion the patient
  Comparison between ID and non ID patients
Occurrence of events (all-cause death, HF-clinically related admissions, CV admissions) | Twelve months after inclusion the patient
  Comparison between ID and non ID patients
Functional Biomarkers (6-minutes walking test [6MWT] distance) | Twelve months after inclusion the patient
  Comparison between ID and non ID patients
Improvement of quality of life using a validated questionnaire (EUROQOL - 5D) | Twelve months after inclusion the patient
  Comparison between ID and non ID patients

CONTACTS AND LOCATIONS:
Overall Officials: Josep Comin Colet, MD, PhD, Principal Investigator — Bellvitge Biomedical Research Institute (IDIBELL) - Hospital Universitari de Bellvitge
Locations (2):
- Spain (2):
  - Hospital Universitari de Bellvtige, L'Hospitalet de Llobregat, Barcelona
  - University Hospital Bellvitge, L'Hospitalet de Llobregat, Barcelona

IPD SHARING:
Plan to Share IPD: No